CLINICAL TRIAL: NCT01011504
Title: A Registry Study to Determine Utilisation Patterns in Patients Receiving Angiox®, and Collect Descriptive Safety and Outcome Data to Inform the Risk Management Strategy for Europe.
Brief Title: Utilisation of Angiox® in European Practice
Acronym: EURO-vision
Status: Completed | Type: Observational
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Other Study IDs: TMC-BIV-08-02
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Stable Angina (SA); NSTE-ACS (NSTEMI and UA); STEMI (STE-ACS)
MeSH Terms: conditions — Angina, Stable; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to determine utilisation patterns in patients receiving Angiox® in participating European centres. Additionally, through the collection of descriptive safety and outcomes data, this study will contribute to the Risk Management strategy for Europe

ELIGIBILITY:
Inclusion Criteria:

* Eligible for, and receive treatment with Angiox®.
* Willing and able to provide written informed consent to the use of their data in accordance with relevant local Data Protection laws, policies and regulations

Exclusion Criteria:

* Participation in other interventional clinical research studies involving the evaluation of investigational drugs, including Angiox®, or devices at the time of enrolment.
* Patients not eligible for treatment for Angiox®.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately, 2,000 patients will be included at centres throughout Europe
Sampling Method: Probability Sample
Enrollment: 2019 (Actual)
Dates: Start 2009-05; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Posology and usage patterns of Angiox®: Dose(s) and time of bolus and infusion administered | from hospital admission until hospital discharge, or 7 days after administration (which ever is earlier).

SECONDARY OUTCOMES:
Death Myocardial infarction Unplanned revascularisation Stroke Major* and minor bleeding Thrombocytopenia Stent thrombosis Adverse events and serious adverse events | measured in-hospital (prior to discharge), and at post-hospital discharge in outpatient as per local practice (30 days)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Nienaber, Prof., Principal Investigator; Martial Hamon, Prof, Principal Investigator
Locations (2):
- Centre Hospitalier Universitaire de Caen, Caen, France
- Medizinische Klinik I Kardiologie/Pneumologie/Internistische, Rostock, Germany